CLINICAL TRIAL: NCT03474640
Title: A Phase 1, Multicenter, Open-label Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of TAB001 in Subjects With Advanced Malignancies
Brief Title: Safety, Tolerability and Pharmacokinetics of an Anti-PD-1 Monoclonal Antibody in Subjects With Advanced Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: TopAlliance Biosciences (Industry)
Collaborators: Shanghai Junshi Bioscience Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TAB001-01
Record Dates: First submitted 2018-02-05; First posted 2018-03-22 (Actual); Results first posted 2024-11-22 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-10

CONDITIONS: Advanced Malignancies
Keywords: immunotherapy; check point inhibitor; PD-1 antibody; solid tumor; esophageal carcinoma; gastric carcinoma; nasopharyngeal carcinoma; hepatocellular carcinoma; soft tissue sarcoma; chondrosarcoma; orphan tumors; phase 1 trial
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms; Nasopharyngeal Carcinoma; Carcinoma, Hepatocellular; Sarcoma; Chondrosarcoma | interventions — toripalimab; Medicare Part B

STUDY DESIGN:
Intervention Model Description: Part A: sequential dose escalation followed by activity estimation in disease specific cohorts at the RP2D.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part A (Experimental): Sequential dose escalation (3+3)
  Interventions: Biological: Part A
- Part B (Experimental): Indication specific dose cohorts: Esophageal Cancer, Gastric Cancer/GEJ, Biliary Tract Cancer, Soft Tissue Sarcoma (excluding Leiomyosarcoma) or Chondrosarcoma, Neuroendocrine Cancer, and other tumors (including Nasopharyngeal Cancer (NPC), Hepatocellular Carcinoma (HCC), MSI-H/dMMR tumors).
  Interventions: Biological: Part B

INTERVENTIONS:
Biological: Part A — Part A: 80, 240, and 480 mg IV every 14 days.
  Other Names: Toripalimab, TAB001, JS001
  Arms: Part A
Biological: Part B — Part B: 240 mg IV every 3 weeks
  Other Names: Toripalimab, TAB001, JS001
  Arms: Part B

SUMMARY:
The primary objective is to assess the safety and tolerability of Toripalimab in subjects with various advanced malignancies and to evaluate the recommended Phase 2 dose.

The secondary objectives are to: 1) describe the pharmacokinetic (PK) profile of Toripalimab, 2) evaluate antitumor activity of Toripalimab; 3) determine the immunogenicity of Toripalimab; 4) evaluate overall survival.

The exploratory objectives are to: 1) evaluate biomarkers that may correlate with activity of Toripalimab, 2) evaluate pharmacodynamic effects of Toripalimab on its target receptor, programmed cell death 1 (PD-1), as well as effects on the immune system. 3) evaluate the utility of PD-L1 & additional exploratory markers as biomarkers that could aid in selection of appropriate subjects for TAB001 therapy, and 4) identification of additional biomarkers correlating with response to treatment with TAB001.

DETAILED DESCRIPTION:
OVERVIEW: This is a Phase 1, open-label, 2-part (Part A = dose-escalation, Part B = multiple disease-specific cohort expansion) study to evaluate the safety, tolerability, PK, immunogenicity, and antitumor activity of toripalimab administered intravenously (IV) every 2 weeks (Q2W) of each 28-day cycle in Part A or 240 mg IV every 3 weeks (Q3W) of each 42-day cycle in Part B in adults with advanced solid tumors with disease progression following standard therapy or for which no standard therapy existed.

Part A used a 3+3 design and enrolled cohorts of 3-6 patients sequentially at escalating doses of 80, 240 an 480 mg Q2W to determine the MTD or MFD and the RP2D; up to 18 patients could be enrolled in the dose-escalation phase. Once a dose-limiting toxicity (DLT) occurred among the first 3 patients, the dose cohort would be expanded to a total of 6 patients. Patients who did not complete the 28-day DLT evaluation period for reasons other than toxicity were to be replaced. Dose escalation was to continue to the highest planned dose level (480 mg) or until identification of the MTD or the MFD. In addition, any cohort that had not exceeded the MTD could be expanded up to a maximum of 10 patients for further evaluation of safety and efficacy. Part A enrollment was limited to immunotherapy-naïve patients (defined as no prior exposure to immunotherapy, including but not limited to, anti-CTLA-4, anti-PD-1, or anti-PD-L1 antibodies; prior use of tumor vaccines was permitted).

In Part B, toripalimab administered at the RP2D, based on Part A, was to be evaluated for safety and antitumor activity. Enrollment was limited to patients who had not received a prior anti-PD-1, anti-PD-L1, or anti-PD-L2 antibody. Up to 280 patients with specified solid tumors could be enrolled in the cohort expansion phase with a maximum of 40 patients to be enrolled in each disease-specific cohort with the exception of the sarcoma cohort, in which a maximum of 80 patients could be enrolled.

The tumor status of all patients was to be evaluated by the investigator according to the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 and the immune-related Response Evaluation Criteria in Solid Tumors (irRECIST). In Part A, radiological assessment of tumor response status was to be performed approximately every 8 weeks (± 10 days) for the first 12 months and approximately every 12 weeks (± 10 days) thereafter, unless the investigator determined it was more appropriate to continue the radiological assessments approximately every 8 weeks. In Part B, radiological assessment of tumor response status was to be performed approximately every 9 weeks (± 10 days) for the first 12 months and approximately every 18 weeks (± 10 days) thereafter, unless the investigator determined it was more appropriate to continue the radiological assessments approximately every 9 weeks.

Patients received toripalimab Q2W (± 2 days) in Part A or Q3W (± 2 days) in Part B, until documentation of confirmed progressive disease (a repeat scan was to be conducted within 4 weeks ± 2 days in Part A and within 6 weeks ± 2 days in Part B to confirm disease progression per irRECIST), unacceptable toxicity, withdrawal of consent, intercurrent illness preventing further administration of toripalimab, or if the investigator considered it in the best interest of the patient to discontinue toripalimab. If feasible, all patients were to be followed for progression-free survival (PFS) and overall survival (OS) (Part B only) until the end of the study.

AEs and serious adverse events (SAEs) were to be captured from the start of the first dose of toripalimab through 90 days after the last dose of toripalimab unless a patient received another experimental or anticancer therapy, in which case only related AEs or SAEs were to be collected through 90 days after the last dose of toripalimab.

Serum samples and tumor tissues were collected for PK, pharmacodynamics, anti-drug antibody (ADA) and biomarkers determination during the study.

ELIGIBILITY:
Inclusion Criteria:

1. Willing to sign Informed Consent;
2. Part A, must have a histologically or cytologically documented, incurable, or metastatic solid tumor that has progressed on, or been intolerant to, all standard systemic therapy options for the tumor type in the metastatic setting, or must have a tumor type for which no such standard systemic option exists;
3. Part B, must have a histologically or cytologically documented diagnosis of esophageal or gastric carcinoma, nasopharyngeal carcinoma (NPC), hepatocellular carcinoma (HCC), both soft tissue sarcoma (excluding leiomyosarcoma), chondrosarcoma, or with agreement of the sponsor, or other tumors who have received at least one line of standard systemic therapy for their respective tumor type in the metastatic setting with progressive locally advanced or metastatic disease that is not amenable to definitive local therapy with curative intent. Patient with MSI-H/dMMR Tumors are eligible to enroll.

   1. Subjects with NPC must have received, or been intolerant to, a platinum-based combination as part of their prior therapy for advanced/metastatic disease;
   2. Subjects with soft tissue sarcoma and chondrosarcoma must have radiographic evidence of progression within the previous 6 months and must have received at least 1 line of systemic therapy;
   3. Subjects with esophageal cancer must have received, or been intolerant to, a platinum-based combination as part of their prior therapy for advanced/metastatic disease;
   4. Subjects with gastric cancer must have received, or been intolerant to, a fluoropyrimidine-platinum combination as part of their prior therapy for advanced/metastatic disease;
   5. Subjects with HCC must have received (or been intolerant to) sorafenib as part of their prior therapy for advanced metastatic disease.
4. Measurable disease per RECIST v1.1 and irRECIST;
5. ECOG performance status of 0 or 1;
6. Adequate organ and marrow function;
7. Willingness to provide consent for biopsy samples;
8. For females of childbearing potential, use effective contraception from time of screening though 90 days post last dose of Toripalimab.

Exclusion Criteria:

1. Concurrent enrollment in another clinical study, unless it is an observational (non-interventional) clinical study or the follow-up period of an interventional study;
2. Any concurrent chemotherapy, radiotherapy, immunotherapy, or biologic therapy for cancer treatment. Concurrent use of hormones for non-cancer related conditions is acceptable (e.g., insulin for diabetes & hormone replacement therapy). Local treatment of isolated lesions for palliative intent is acceptable;
3. Receipt of any investigational anti-cancer therapy within 4 weeks prior to first dose of Toripalimab;
4. Current use or prior use of immunosuppressive medication within 4 weeks prior to first dose of Toripalimab, with the exception of intranasal and inhaled corticosteroids or systemic corticosteroids not to exceed 10mg/day of prednisone or equivalent;
5. Part A: Prior exposure to immunotherapy such as but not limited to other anti-CTLA- 4, anti-PD-1, or anti-PD-L1 antibodies excluding vaccines. Part B: Exclusion of prior immunotherapy exposure will be limited to anti-PD-1, anti-PD-L1, or anti-PD-L2;
6. Prior allogeneic bone marrow transplantation or prior solid organ transplantation;
7. Major surgery within 4 weeks prior to first dose of Toripalimab or still recovering from prior surgery;
8. Unresolved toxicities from prior anticancer therapy defined as having not resolved to baseline or to Grade 0 or 1, or to levels dictated in the inclusion/exclusion criteria with the exception of alopecia;
9. Active or prior documented autoimmune disease within the past 2 years. Subjects with vitiligo, Grave's disease, or psoriasis not requiring systemic treatment within the past 2 years are not excluded;
10. Known history of tuberculosis;
11. Known to be human immunodeficiency virus (HIV) positive, hepatitis B, or hepatitis C positive;
12. Active or prior documented inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis);
13. History of primary immunodeficiency;
14. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure according to NYHA Functional Classification ≥3, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, active peptic ulcer disease or gastritis, or psychiatric illness/social situations that would limit compliance with study requirements, substantially increase risk of incurring adverse events from Toripalimab, or compromise the ability of the subject to give written informed consent;
15. Symptomatic or untreated central nervous system metastases requiring concurrent treatment, inclusive of but not limited to surgery, radiation, and/or corticosteroids. Subjects with previously treated brain metastases may participate provided they are clinically stable for at least 4 weeks prior to study entry, have no evidence of new or enlarging metastases, and are off steroids;
16. Receipt of live attenuated vaccination within 30 days prior to study entry or within 4 weeks of receiving Toripalimab;
17. Pregnancy or breastfeeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2018-02-21 (Actual); Primary Completion 2022-06-07 (Actual); Study Completion 2022-07-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sheng Yao, PhD, Study Director — TopAlliance Biosciences, Inc.
Locations (14):
- United States (14):
  - Sarcoma Oncology Research Center, Santa Monica, California
  - University of Colorado Denver, Aurora, Colorado
  - University of Miami Hospital Sylvester Comprehensive Cancer Center, Miami, Florida
  - Florida Cancer Specialists, Sarasota, Florida
  - University of Maryland Marlene and Stewart Greenebaum Comprehensive Cancer Center, Baltimore, Maryland
  - Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - Karmanos Cancer Institute, Detroit, Michigan
  - Mayo Clinic-Rochester, Rochester, Minnesota
  - Carolina BioOncology Institute, Huntersville, North Carolina
  - University Hospitals Seidman Cancer Center, Cleveland, Ohio
  - Rhode Island Hospital, Providence, Rhode Island
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Derived] Naing A, Mahipal A, Javle M, Wang J, Bauer TM, Bajor DL, Elias AD, Shields A, Davis E, Chawla S, Safran H, Powderly JD, D'Amato G, Meyer CF, Tang X, Yao S, Keegan P. Safety and Efficacy of Toripalimab in Patients with Cholangiocarcinoma: An Open-Label, Phase 1 Study. J Immunother Precis Oncol. 2025 Jan 15;8(1):71-81. doi: 10.36401/JIPO-24-8. eCollection 2025 Feb. PMID 39816916

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was initiated on 21 February 2018 (first patient signed the informed consent form) and completed on 07 June 2022. This study was conducted and screened patients in 14 sites in the United States.
Pre-assignment Details: Once a patient was determined to be eligible, the patient was considered "enrolled" and an identification number was to be assigned, which denoted the dose-level or disease-specific cohort assignment.
  Patients who failed to meet the inclusion/exclusion criteria (i.e., screen failures) might be rescreened up to 3 times and would maintain their same screening number. Study participation began once a patient received the first dose of toripalimab.
Groups:
- Toripalimab 80 mg Repeat Dose Every 14 Days: 3-6 subjects (Part A) Toripalimab 80 mg repeat dose every 14 days
- Toripalimab 240 mg Repeat Dose Every 14 Days: 3-6 subjects (Part A) Toripalimab 240 mg repeat dose every 14 days
- Toripalimab 480 mg Repeat Dose Every 14 Days: 3-6 subjects (Part A) Toripalimab 480 mg repeat dose every 14 days
- Biliary Tract Cancer: Toripalimab 240 mg IV every 3 weeks
  42 patients
- Sarcoma: Toripalimab 240 mg IV every 3 weeks
  59 patients
- Esophageal Cancer: Toripalimab 240 mg IV every 3 weeks
  11 patients
- Gastric Cancer: Toripalimab 240 mg IV every 3 weeks
  29 patients
- Neuroendocrine Cancer: Toripalimab 240 mg IV every 3 weeks
  22 patients
- Other Tumors: Toripalimab 240 mg IV every 3 weeks
  3 patients
Period: Overall Study
Arm/Group | Toripalimab 80 mg Repeat Dose Every 14 Days | Toripalimab 240 mg Repeat Dose Every 14 Days | Toripalimab 480 mg Repeat Dose Every 14 Days | Biliary Tract Cancer | Sarcoma | Esophageal Cancer | Gastric Cancer | Neuroendocrine Cancer | Other Tumors
Started | 3 | 8 | 7 | 42 | 59 | 11 | 29 | 22 | 3
Completed | 0 | 0 | 2 | 8 | 7 | 1 | 3 | 6 | 1
Not Completed | 3 | 8 | 5 | 34 | 52 | 10 | 26 | 16 | 2

BASELINE CHARACTERISTICS:
Groups:
- Part A: Toripalimab 80 mg Every 14 Days; Part A: Toripalimab 240 mg Every 14 Days; Part A: Toripalimab 480 mg Every 14 Days: 3-6 subjects (Part A)
  Patients with relapsed or refractory solid tumors who have progressed on standard treatment
- Part B: Sarcoma: 44-80 subjects (Part B) soft tissue sarcoma (excluding leiomyosarcoma) or chondrosarcoma who have progressed on at least one prior regimen for metastatic disease
  Toripalimab, 240 mg IV every 21 days
- Part B: Other Tumors: 22-40 subjects (Part B) nasopharyngeal cancer (NPC), hepatocellular cancer (HCC),MSI-H/dMMR who have progressed on at least one prior regimen for metastatic disease
  Toripalimab, 240 mg IV every 21 days
- Part B: Esophogeal: 22-40 subjects (Part B) esophogeal cancer who have progressed on at least one prior regimen for metastatic disease
  Toripalimab, 240 mg IV every 21 days
- Part B: Gastric/GEJ: 22-40 subjects (Part B) gastric/GEJ cancer who have progressed on at least one prior regimen for metastatic disease
  Toripalimab, 240 mg IV every 21 days
- Part B: Biliary Tract: 22-40 subjects (Part B) biliary tract cancer who have progressed on at least one prior regimen for metastatic disease
  Toripalimab, 240 mg IV every 21 day
- Part B: Neuroendocrine: 22-40 subjects (Part B) neuroendocrine cancer who have progressed on at least one prior regimen for metastatic disease
  Toripalimab, 240 mg IV every 21 day
- Total: Total of all reporting groups
Arm/Group | Part A: Toripalimab 80 mg Every 14 Days | Part A: Toripalimab 240 mg Every 14 Days | Part A: Toripalimab 480 mg Every 14 Days | Part B: Sarcoma | Part B: Other Tumors | Part B: Esophogeal | Part B: Gastric/GEJ | Part B: Biliary Tract | Part B: Neuroendocrine | Total
Number analyzed (Participants) | 3 | 8 | 7 | 59 | 3 | 11 | 29 | 42 | 22 | 184
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 6 | 5 | 37 | 2 | 6 | 11 | 25 | 9 | 103
  >=65 years | 1 | 2 | 2 | 22 | 1 | 5 | 18 | 17 | 13 | 81
Age, Continuous [Median (Full Range); unit: years] | 62 [62 to 69] | 60.5 [29 to 66] | 55 [46 to 73] | 60 [21 to 85] | 40 [38 to 75] | 63 [53 to 78] | 66 [29 to 83] | 60.5 [35 to 85] | 65.5 [34 to 84] | 62 [21 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 5 | 5 | 26 | 1 | 2 | 8 | 28 | 4 | 80
  Male | 2 | 3 | 2 | 33 | 2 | 9 | 21 | 14 | 18 | 104
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 7 | 2 | 1 | 1 | 1 | 1 | 14
  Not Hispanic or Latino | 3 | 7 | 7 | 49 | 1 | 9 | 28 | 40 | 20 | 164
  Unknown or Not Reported | 0 | 0 | 0 | 3 | 0 | 1 | 0 | 1 | 1 | 6
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 8 | 7 | 59 | 3 | 11 | 29 | 42 | 22 | 184

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-related Adverse Events as Assessed by CTCAE v4.0
Description: To assess the number of treatment-related adverse events in the toripalimab arm as assessed by CTCAE v4.0
Time Frame: Through study completion, an estimated period of approximately 2 years.
Measure: Count of Participants; unit: Participants
Groups:
- Part A: 80 mg: Part A 80 mg IV toripalimab every 14 days Sequential dose escalation (3+3)
- Part A: 240 mg: Part A 240 mg IV toripalimab every 14 days Sequential dose escalation (3+3)
- Part A: 480 mg: Part A 480 mg IV toripalimab every 14 days Sequential dose escalation (3+3)
- Part B: Sarcoma: 44-80 subjects (Part B) soft tissue sarcoma (excluding leiomyosarcoma or chondrosarcoma) who have progressed on at least one prior therapy regimen for metastatic disease. Toripalimab 240 mg IV every 21 days.
- Part B: Other Tumors: 22-40 subjects (Part B)nasopharyngeal cancer (NPC), hepatocellular cancer (HCC),MSI-H/dMMR who have progressed on at least one prior regimen for metastatic disease. Toripalimab 240 mg IV every 21 days.
- Part B: Esophageal: 22-40 subjects (PartB) esophogeal cancer who have progressed on at least one prior regimen for metastatic disease. Toripalimab 240 mg IV every 21days.
- Part B: Gastric/GEJ: 22-40 subjects (PartB) gastric/GEJ cancer who have progressed on at least one prior regimen for metastatic disease. Toripalimab,240 mg IV every 21days.
- Part B: Biliary Tract: 22-40 subjects (PartB) biliary tract cancer who have progressed on at least one prior regimen for metastatic disease. Toripalimab,240 mg IV every 21 days.
- Part B: Neuroendocrine: 22-40 subjects (Part B)neuroendocrine cancer who have progressed on at least one prior regimen for metastatic disease.
  Toripalimab 240 mg IV every 21 days.
Arm/Group | Part A: 80 mg | Part A: 240 mg | Part A: 480 mg | Part B: Sarcoma | Part B: Other Tumors | Part B: Esophageal | Part B: Gastric/GEJ | Part B: Biliary Tract | Part B: Neuroendocrine
Number analyzed (Participants) | 3 | 8 | 7 | 59 | 3 | 11 | 29 | 42 | 22
Participants | 2 | 5 | 5 | 33 | 2 | 7 | 15 | 27 | 14

2. Secondary Outcome: Objective Response Rate (ORR)
Description: The treatment effect of Toripalimab was assessed using RECIST 1.1 to determine objective response rate. ORR was defined and analyzed as the number of subjects achieving BOR of CR or PR, divided by the number of treated subjects.
  Subjects without at least one post-baseline radiological assessment were treated as non-responders. ORR was presented by dose cohort in Part A and tumor type in Part B, with 95% confidence intervals.
Time Frame: Every 8 weeks (Part A) or every 9 weeks (Part B) through study completion, an estimated duration of 2 years.
Measure: Count of Participants; unit: Participants
Groups:
- Part A: 80 mg: Part A 80 mg IV toripalimab every 14 days
- Part A: 240 mg: Part A 240 mg IV toripalimab every 14 days
- Part A: 480 mg: Part A 480 mg IV toripalimab every 14 days
- Part B: Sarcoma: 44-80 subjects(Part B) soft tissue sarcoma (excluding leiomyosarcoma or chondrosarcoma)who have progressed on at least one prior regimen for metastatic disease.
  Toripalimab 240 mg IV for 21 days.
- Part B: Other Tumors: 22-40 subjects (Part B) nasopharyngeal cancer (NPC), hepatocellular cancer (HCC),MSI-H/dMMR who have progressed on at least one prior regimen for metastatic disease.
  Toripalimab 240 mg IV every 21 days.
- Part B: Esophageal: 22-40 subjects (Part B) esophogeal cancer who have progressed on at least one prior regimen for metastatic disease.
  Toripalimab 240 mg IV every 21days.
- Part B: Gastric/GEJ: 22-40 subjects (Part B) gastric/GEJ cancer who have progressed on at least one prior regimen for metastatic disease.
  Toripalimab 240 mg IV every 21days.
- Part B: Biliary Tract: 22-40 subjects (Part B) biliary tract cancer who have progressed on at least one prior regimen for metastatic disease.
  Toripalimab 240 mg IV every 21 days.
- Part B: Neuroendocrine: 22-40 subjects (Part B) neuroendocrine cancer who have progressed on at least one prior regimen for metastatic disease. Toripalimab 240 mg IV every 21 days.
Arm/Group | Part A: 80 mg | Part A: 240 mg | Part A: 480 mg | Part B: Sarcoma | Part B: Other Tumors | Part B: Esophageal | Part B: Gastric/GEJ | Part B: Biliary Tract | Part B: Neuroendocrine
Number analyzed (Participants) | 3 | 8 | 7 | 59 | 3 | 11 | 29 | 42 | 22
Participants | 0 | 0 | 0 | 5 | 0 | 3 | 1 | 2 | 3

3. Secondary Outcome: Disease Control Rate (DCR)
Description: The treatment effect of Toripalimab was assessed using RECIST 1.1 to determine objective response rate. ORR was defined and analyzed as the number of subjects achieving BOR of CR, PR, or SD divided by the number of treated subjects.
  Subjects without at least one post-baseline radiological assessment were treated as non-responders. DCR was presented by dose cohort in Part A and tumor type in Part B, with 95% confidence intervals.
Time Frame: Every 8 weeks (Part A) or every 9 weeks (Part B) through study completion, an estimated duration of 2 years.
Measure: Count of Participants; unit: Participants
Groups:
- Part B: Sarcoma: 44-80 subjects (Part B) soft tissue sarcoma(excluding leiomyosarcoma or chondrosarcoma) who have progressed on at least one prior regimen for metastatic disease. Toripalimab 240mg IV every 21days.
- Part B: Other Tumors: 22-40 subjects (Part B) nasopharyngeal cancer (NPC),hepatocellularcancer (HCC), MSI-H/dMMR who have progressed on at least one prior regimen for metastatic disease. Toripalimab 240 mg IV every 21 days.
- Part B: Esophageal Tumors: 22-40 subjects (Part B) esophogeal cancer who have progressed on at least one prior regimen for metastatic disease.
  Toripalimab 240 mg IV every 21days.
Arm/Group | Part A: 80 mg | Part A: 240 mg | Part A: 480 mg | Part B: Sarcoma | Part B: Other Tumors | Part B: Esophageal Tumors | Part B: Gastric/GEJ | Part B: Biliary Tract | Part B: Neuroendocrine
Number analyzed (Participants) | 3 | 8 | 7 | 59 | 3 | 11 | 29 | 42 | 22
Participants | 0 | 5 | 6 | 25 | 1 | 4 | 7 | 17 | 11

4. Secondary Outcome: Progression-Free Survival (PFS)
Description: The treatment effect of Toripalimab was assessed using RECIST 1.1 to determine progression-free survival time. PFS was defined as the time from the first dose of toripalimab to the first PD or death due to any cause, whichever occurred first and was analyzed separately for each cohort in Part B only,
Time Frame: Every 8 weeks (Part A) or every 9 weeks (Part B) through study completion, an estimated duration of 2 years.
Measure: Median (Inter-Quartile Range); unit: months
Groups:
- Part B: Sarcoma: Part B Sarcoma: 240 mg toripalimab IV every 3 weeks
- Part B: Other Tumors: Part B Other Tumors: 240 mg toripalimab IV every 3 weeks
- Part B: Esophageal: Part B Esophageal: 240 mg toripalimab IV every 3 weeks
- Part B: Gastric/GEJ: Part B Gastric/GEJ: 240 mg toripalimab IV every 3 weeks
- Part B: Biliary Tract: Part B Biliary Tract: 240 mg toripalimab IV every 3 weeks
- Part B: Neuroendocrine: Part B Neuroendocrine: 240 mg toripalimab IV every 3 weeks
Arm/Group | Part B: Sarcoma | Part B: Other Tumors | Part B: Esophageal | Part B: Gastric/GEJ | Part B: Biliary Tract | Part B: Neuroendocrine
Number analyzed (Participants) | 59 | 3 | 11 | 29 | 42 | 22
months | 2.2 [1.8 to 6.2] | 1.4 [1.0 to 4.1] | 2.1 [2.1 to 6.2] | 2.1 [1.5 to 4.0] | 2.1 [1.8 to 4.1] | 6.4 [1.5 to NA] — NA, N.E.= Not Estimable, insufficient number of patients with events

5. Secondary Outcome: Overall Survival (OS)
Description: The treatment effect of Toripalimab was assessed using RECIST 1.1 to determine overall survival (OS) analysis by tumor type in Part B. OS was defined as the time from date the first dose of toripalimab until death due to any cause. OS time for subjects not achieving the endpoint was censored at the last known alive date.
Time Frame: Through study completion, an estimated duration of 2 years.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part B: Sarcoma | Part B: Other Tumors | Part B: Esophageal | Part B: Gastric/GEJ | Part B: Biliary Tract | Part B: Neuroendocrine
Number analyzed (Participants) | 59 | 3 | 11 | 29 | 42 | 22
months | 4.9 [3.71 to 6.54] | 1.4 [1.12 to NA] — NA, N.E.= Not Estimable, insufficient number of patients with events | 5.7 [0.79 to 21.72] | 3.5 [2.33 to 6.93] | 4.4 [3.48 to 4.86] | 4.2 [2.60 to 8.25]

ADVERSE EVENTS:
Time Frame: All the TEAEs from first dose to 90 days after the last dose of toripalimab were included in the safety evaluation, an average duration of six months, up to two years.
Description: Safety data are based on the June 7, 2022 data cut-off date.
Groups:
- Toripalimab 80 mg Every 14 Days; Toripalimab 240 mg Every 14 Days; Toripalimab 480 mg Every 14 Days: 3-6 subjects (Part A)
  Patients with relapsed or refractory solid tumors who have progressed on standard treatment
- Sarcoma: 44-80 subjects (Part B) soft tissue sarcoma (excluding leiomyosarcoma) or chondrosarcoma who have progressed on at least one prior regimen for metastatic disease
  Toripalimab, 240 mg IV every 21 days
- Other Tumors: 22-40 subjects (Part B) nasopharyngeal cancer (NPC), hepatocellular cancer (HCC),MSI-H/dMMR who have progressed on at least one prior regimen for metastatic disease
  Toripalimab, 240 mg IV every 21 days
- Esophogeal: 22-40 subjects (Part B) esophogeal cancer who have progressed on at least one prior regimen for metastatic disease
  Toripalimab, 240 mg IV every 21 days
- Gastric/GEJ: 22-40 subjects (Part B) gastric/GEJ cancer who have progressed on at least one prior regimen for metastatic disease
  Toripalimab, 240 mg IV every 21 days
- Biliary Tract: 22-40 subjects (Part B) biliary tract cancer who have progressed on at least one prior regimen for metastatic disease
  Toripalimab, 240 mg IV every 21 day
- Neuroendocrine: 22-40 subjects (Part B) neuroendocrine cancer who have progressed on at least one prior regimen for metastatic disease
  Toripalimab, 240 mg IV every 21 day
Arm/Group | Toripalimab 80 mg Every 14 Days | Toripalimab 240 mg Every 14 Days | Toripalimab 480 mg Every 14 Days | Sarcoma | Other Tumors | Esophogeal | Gastric/GEJ | Biliary Tract | Neuroendocrine
All-Cause Mortality (participants affected / at risk) | 1/3 | 2/8 | 0/7 | 12/59 | 0/3 | 2/11 | 9/29 | 12/42 | 3/22
Serious Adverse Events (participants affected / at risk) | 2/3 | 2/8 | 4/7 | 23/59 | 1/3 | 3/11 | 11/29 | 23/42 | 6/22
Other Adverse Events (participants affected / at risk) | 2/3 | 5/8 | 5/7 | 33/59 | 2/3 | 7/11 | 15/29 | 27/42 | 14/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Toripalimab 80 mg Every 14 Days (N=3) | Toripalimab 240 mg Every 14 Days (N=8) | Toripalimab 480 mg Every 14 Days (N=7) | Sarcoma (N=59) | Other Tumors (N=3) | Esophogeal (N=11) | Gastric/GEJ (N=29) | Biliary Tract (N=42) | Neuroendocrine (N=22)
Gastrointestinal Disorders (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 6 | 5 | 1
Infections and Infestations (Infections and infestations) | 0 | 0 | 1 | 4 | 0 | 2 | 1 | 8 | 0
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 7 | 0 | 0 | 5 | 2 | 0
Metabolism and Nutrition Disorders (Metabolism and nutrition disorders) | 0 | 0 | 1 | 3 | 1 | 0 | 2 | 1 | 2
Nervous System Disorders (Nervous system disorders) | 1 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0
Musculoskeletal and Connective Tissue Disorders (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Reproductive System and Breast Disorders (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal and Urinary Disorders (Renal and urinary disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 3 | 1
General Disorders (General disorders) | 0 | 0 | 0 | 3 | 0 | 0 | 1 | 1 | 2
Vascular Disorders (Vascular disorders) | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0
Hepatobiliary Disorders (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Injury, Poisoning and Procedural Complications (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 1
Blood and Lymphatic System Disorders (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cardiac Disorders (Cardiac disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Skin and Subcutaneous Disorders (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Endocrine Disorders (Endocrine disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Immune System Disorders (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Toripalimab 80 mg Every 14 Days (N=3) | Toripalimab 240 mg Every 14 Days (N=8) | Toripalimab 480 mg Every 14 Days (N=7) | Sarcoma (N=59) | Other Tumors (N=3) | Esophogeal (N=11) | Gastric/GEJ (N=29) | Biliary Tract (N=42) | Neuroendocrine (N=22)
Skin and Subcutaneous Disorder (Skin and subcutaneous tissue disorders) | 0 | 2 | 2 | 9 | 2 | 0 | 6 | 2 | 5 — Pruritus, dry skin
Investigations (Investigations) | 1 | 0 | 1 | 12 | 0 | 3 | 4 | 12 | 3 — transaminases increased, lipases increased
General Disorders (General disorders) | 0 | 2 | 1 | 10 | 0 | 3 | 4 | 11 | 6 — Fatigue, chills, oedema
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 0 | 1 | 1 | 5 | 0 | 2 | 4 | 4 | 2 — Decreased appetite
Gastrointestinal Disorders (Gastrointestinal disorders) | 0 | 2 | 1 | 10 | 0 | 3 | 4 | 11 | 4 — Diarrhea, nausea, abdominal pain
Blood and Lymphatic Disorders (Blood and lymphatic system disorders) | 1 | 3 | 1 | 5 | 0 | 0 | 2 | 6 | 1 — Lymphopenia, anemia, leukopenia, neutropenia, pancytopenia, thrombocytopenia
Endocrine Disorders (Endocrine disorders) | 0 | 1 | 0 | 10 | 1 | 2 | 1 | 1 | 2 — Hyperthyroidism, hypothyroidism
Nervous System Disorders (Nervous system disorders) | 1 | 1 | 0 | 1 | 0 | 1 | 5 | 1 | 0 — Headache, peripheral neuropathy, dizziness, dysgeusia
Musculoskeletal and Connective Tissue Disorders (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 4 | 1 — Musculoskeletal pain, muscular weakness
Injury, Poisoning, and Procedural Complications (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 1 — Infusion related reaction
Cardiac Disorders (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 — Myocarditis
Vascular Disorders (Vascular disorders) | 0 | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 0 — Hypotension
Neoplasms benign, malignant, and unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 — Tumor pain
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-06-25): https://cdn.clinicaltrials.gov/large-docs/40/NCT03474640/Prot_000.pdf
  • Statistical Analysis Plan (2022-07-21): https://cdn.clinicaltrials.gov/large-docs/40/NCT03474640/SAP_001.pdf